CLINICAL TRIAL: NCT01015196
Title: AML 2001: a Phase III Prospective Randomized Study Comparing One or Two High Dose Chemotherapy Regimen Followed by Autologous Stem Cell Transplantation (ASCT) as Consolidation Strategy for Adults Aged 15 to 60 With Acute Myeloid Leukemia (AML) in First Complete Remission (CR).rémission complète d'Une Leucémie Aiguë Myéloblastique
Brief Title: Prospective Randomized Study Comparing One or Two High Dose Chemotherapy Regimen Followed by Autologous Stem Cell Transplantation
Acronym: AML2001
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Cellule de promotion de la recherche clinique, Nantes University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD 99/10-L
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia in first complete remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Idarubicine (Active Comparator)
  Interventions: Drug: Zavedos
- Daunorubicine (Experimental)
  Interventions: Drug: Cerubidine

INTERVENTIONS:
Drug: Zavedos
  Arms: Idarubicine
Drug: Cerubidine
  Arms: Daunorubicine

SUMMARY:
First randomization:

After inclusion Use of Daunorubicin (arm D) or Idarubicin (arm I) as anthracyclin during all courses of chemotherapy (induction, consolidation courses before ASCT)

Second randomization:

After achieving 1st CR: all patients received non intensive consolidation course Familial HLA typing required for all patients

Patients with HLA-identical sibling:

Patients with very good prognostic factors (CBF leukemias, WBC < 30 giga/l at diagnosis, 1st CR after one induction course) = arm C: no allogeneic stem cell transplantation in 1st CR; received 2 more courses of intensive consolidation chemotherapy All others patients received an allogeneic transplant For patients aged less than 51 = arm M: upfront myeloablative conditioning regimen For patients aged over 51 and less than 61= arm m: intensive chemotherapy consolidation course.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 to 60 years
* Diagnosis untreated AML (FAB 0 to 2, 4 to 7): more than 20% marrow blasts according to WHO classification
* Signed informed consent required

Exclusion Criteria:

* AML3 subtype
* Previous diagnosis of myelodysplastic syndrome (MDS) or myeloproliferative disease; patients with previous chemotherapy or radiotherapy were eligible if they had no previous diagnosis of MDS
* Isolated extramedullary disease
* Inadequate performance status (≥ 3), cardiac function (LVEF < 40%, severe arythmia or unstable coronary disease), renal function (creatininine > 150 µmol/l), liver functional tests (bilirubin > 35 µmol/l, liver enzymes > 4 times normal values); life expectancy < 3 months
* Informed consent refusal

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 832 (Actual)
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Bertoli S, Bories P, Bene MC, Daliphard S, Lioure B, Pigneux A, Vey N, Delaunay J, Leymarie V, Luquet I, Blanchet O, Cornillet-Lefebvre P, Hunault M, Bouscary D, Fegueux N, Guardiola P, Dreyfus F, Harousseau JL, Cahn JY, Ifrah N, Recher C; Groupe Ouest-Est d'Etude des Leucemies Aigues et Autres Maladies du Sang (GOELAMS). Prognostic impact of day 15 blast clearance in risk-adapted remission induction chemotherapy for younger patients with acute myeloid leukemia: long-term results of the multicenter prospective LAM-2001 trial by the GOELAMS study group. Haematologica. 2014 Jan;99(1):46-53. doi: 10.3324/haematol.2013.091819. Epub 2013 Aug 23. PMID 23975179
- [Derived] Guieze R, Cornillet-Lefebvre P, Lioure B, Blanchet O, Pigneux A, Recher C, Bonmati C, Fegueux N, Bulabois CE, Bouscary D, Vey N, Delain M, Turlure P, Himberlin C, Harousseau JL, Dreyfus F, Bene MC, Ifrah N, Chevallier P; GOELAMS. Role of autologous hematopoietic stem cell transplantation according to the NPM1/FLT3-ITD molecular status for cytogenetically normal AML patients: a GOELAMS study. Am J Hematol. 2012 Dec;87(12):1052-6. doi: 10.1002/ajh.23311. Epub 2012 Aug 22. PMID 22911473
- [Derived] Lioure B, Bene MC, Pigneux A, Huynh A, Chevallier P, Fegueux N, Blaise D, Witz B, Delain M, Cornillon J, Luquet I, Blanchet O, Cornillet-Lefebvre P, Carre M, Hunault M, Larosa F, Lamy T, Randriamalala E, Ojeda-Uribe M, Berthou C, Fornecker L, Harousseau JL, Bouscary D, Ifrah N, Cahn JY; GOELAMS. Early matched sibling hematopoietic cell transplantation for adult AML in first remission using an age-adapted strategy: long-term results of a prospective GOELAMS study. Blood. 2012 Mar 22;119(12):2943-8. doi: 10.1182/blood-2011-05-352989. Epub 2012 Feb 9. PMID 22323482